CLINICAL TRIAL: NCT01582659
Title: Outpatient Treatment of Constipation in Children - a Randomized Interventions Study
Brief Title: Outpatient Treatment of Constipation in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Line Modin (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Sponsor-Investigator, Line Modin, Medical doctor, Vejle Hospital
Organization: Vejle Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OutCon
Record Dates: First submitted 2012-03-27; First posted 2012-04-20 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Constipation
Keywords: constipation; children; outpatient
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- No ekstra counseling (No Intervention): Standardized information about childhood constipation is given and the child receives PEG 3350. No additional follow up appointments are made.
- 2 counseling sessions (Active Comparator): Standardized information about childhood constipation is given and the child receives PEG 3350. 2 additional follow up appointments by telephone are made.
  Interventions: Other: Telephone counseling
- Web access (Active Comparator): Standardized information about childhood constipation is given and the child receives PEG 3350. No additional follow up appointments are made but the family are given access to a website with information about childhood constipation.
  Interventions: Other: Web access

INTERVENTIONS:
Other: Telephone counseling — 2 planned telephone counseling sessions are conducted.
  Other Names: Telephone
  Arms: 2 counseling sessions
Other: Web access — Access to a web site with information about childhood constipation similar to the information given at the first visit to the clinic.
  Other Names: Web
  Arms: Web access

SUMMARY:
Constipation is a condition often seen in children. Constipation is often associated with impaired quality of life of the child and of great concern among parents. Despite the fact that both diagnosis and treatment is a simple task, it is often seen that the treatment fails, and many children are referred to a pediatric ward for specialized treatment.

There is currently little research on the subject and treatment is therefore based on expert knowledge rather than scientific research.

The study objective is to identify the most effective and least stressful treatment of children with constipation for both families and the health care system.

The following will be tested:

Does treatment of constipation in children require specialized knowledge and extensive resources or can the treatment be simplified?

The results from this study are expected to form the basis for a evidence based treatment of children with constipation.

ELIGIBILITY:
Inclusion Criteria:

* Children between 2 and 16 years and referral to our out patient clinic with either constipation or fecal incontinence.
* Patients must fulfill the Rome III criteria of constipation, which mean they must have at least 2 of the following characteristics: fewer than 3 bowel movements weekly, more than 1 episode of fecal incontinence weekly, large stools in the rectum by digital rectal examination or palpable on abdominal examination, occasional passing of large stools, display of retentive posturing and withholding behavior, and painful defecation.

Exclusion Criteria:

* Children with known organic causes of constipation, including Hirschsprungs disease, spinal and anal congenital abnormalities, previous surgery on the colon, inflammatory bowel disease, allergy and metabolic or endocrine diseases.
* Children receiving drugs known to affect bowel function during a 2 month period before initiation.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 239 (Actual)
Dates: Start 2012-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Treatment recovery | 1 year
  Recovery is defined as the child having no symptoms of constipation according to the Rome III chriteria.

SECONDARY OUTCOMES:
Usage of laxative. | 1 year
  Amount of laxative used during the study periode.
Telephone contacts | 1 year
  Number of telephone contacts during the study periode, both planned and unplanned contacts will be noted.

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Jakobsen, MD, PhD, Study Director — Kolding; Poul Erik Kofoed, MD. PHD, Study Chair — Kolding; Line Modin, MD, Principal Investigator — Kolding
Locations (2):
- Denmark (2):
  - Line Modin, Kolding
  - Pediatric department, Kolding Hospital, Kolding

REFERENCES:
- [Derived] Modin L, Walsted AM, Rittig CS, Hansen AV, Jakobsen MS. Follow-up in Childhood Functional Constipation: A Randomized, Controlled Clinical Trial. J Pediatr Gastroenterol Nutr. 2016 Apr;62(4):594-9. doi: 10.1097/MPG.0000000000000974. PMID 26348685